CLINICAL TRIAL: NCT05924581
Title: Validation of Clinical Assessment of Spinal Stiffness in Hyperkyphosis and Scoliosis During Growth
Brief Title: Validation of Clinical Assessment of Spinal Stiffness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ClinTest-HKS
Record Dates: First submitted 2023-06-15; First posted 2023-06-29 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hyperkyphosis; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical assessment of spinal stiffness (Experimental): Patients' back flexibility will be assessed during the medical examination or physiotherapy session through one of the following non-invasive tests:
  * Thoracic Stiffness Test (TST)
  * Scoliosis stiffness test (SST)
  * Kyphosis Stiffness Test (KST) Each test will be carried out at the beginning of the visit and repeated at the end 2 times by different operators, or once by the same operator to verify that the measurements taken at different times are reliable and that the measurements taken by two different operators are reliable.
  Interventions: Other: Clinical assessment of spinal stiffness

INTERVENTIONS:
Other: Clinical assessment of spinal stiffness — The clinical stiffness tests will be applied twice to the same patient by the same operator to verify intra-operator variability and twice by two operators at the same time to verify inter-operator variability.
  The verification of diagnostic accuracy with respect to the radiographic reference standard will be carried out retrospectively by using the data already available and systematically collected in electronic format during medical visits and physiotherapy sessions.

SUMMARY:
This study aims to validate and verify the reliability of the clinical measures used in the daily routine by doctors and therapists that allow assessing the spinal stiffness in all spatial planes. The secondary objective is the verification of the diagnostic accuracy of the most reliable tests in identifying the subjects at risk of failure, using as a radiographic standard the examinations performed by the patients during the treatment (data retrieved retrospectively) using as a control group those patients who did not obtain a correction of the spine curvature.

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis > 10°Cobb or Hyperkyophosis >50° Cobb
* Age between 10 and 17 years old
* Risser between 0 and 5

Exclusion Criteria:

* History of spinal surgery
* Presence of back pain
* Diagnosis of congenital scoliosis or scoliosis secondary to neurological or muscular diseases

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Reliability | through study completion, an average of 6 months
  Test-retest reliability of the three stiffness assessment tests. Inter class correlation will be calculated
Repeatability | through study completion, an average of 6 months
  Inter-Rater and Intra-Rater Repeatability of the three stiffness assessment tests
Diagnostic accuracy | through study completion, an average of 6 months
  diagnostic sensitivity and specificity of each test

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be deposited in an online repository